CLINICAL TRIAL: NCT02565329
Title: Serum Lactate Trend in Liver Resection With Intermittent Pringle Maneuver: The "Square-Root" Shape
Brief Title: Serum Lactate Trend in Liver Resection
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Prof Guido Torzilli, MD, PhD, FACS, University of Milan
Other Study IDs: LacClearance
Record Dates: First submitted 2015-09-23; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Lactase Persistence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aimed to evaluate the correlation between the serum lactate concentration ed cumulative Pringle time after liver resection. In addition, the correlation between lactate clearance and clamping time was investigated.

DETAILED DESCRIPTION:
During liver resection high serum lactate (sLac) concentration can be related to several clinical factors: impairment in lactate metabolism (i.e. extraction and utilization by the liver) or overproduction by splanchnic tissues; restrictive fluid regimen in order to limit the intraoperative back-flow bleeding; ischemia-reperfusion syndrome. However, the Pringle maneuver (temporary clamping of the hepatic hilum) seems having a sensible effect in inducing a significant increase in sLac levels during liver resection, particularly in the event of compromised liver function such as in cirrhosis.

Although the peak of sLac concentration may correlate with outcome, the lactate clearance (cLac) seems to be a better predictor. To date, this relationship has been mainly demonstrated in severe sepsis and shock septic. However, the effective correlation between the cumulative clamping time and cLac has not been clearly investigated. The correlation between cumulative hepatic ischemic time and sLac trend in the perioperative period after liver resection with intermittent PM was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for liver resection for hepatic tumors

Exclusion Criteria:

* Patients who received blood transfusion or affected by chronic renal failure were excluded

Ages: 34 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 133 consecutive patients scheduled for liver resection for primary and secondary tumors
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Serum lactate concentration trend after liver resection | within the first 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guido Guido, Guido, Principal Investigator — Humanitas Research Hospital, Humanitas University, via Manzoni 56, 20089 Milan
Locations (1):
- Department of Hepatobiliary and General Surgery, Humanitas Research Hospital, University of Milan, Rozzano, Milan, Italy